CLINICAL TRIAL: NCT05833568
Title: Double-blind Randomized Controlled Trial of a 10-Hz Transcranial Alternating Current Stimulation to Modulate Brain Activity in Brain-injured Patients With Disorders of Consciousness
Brief Title: Five-day 20-minute 10-Hz tACS in Patients With a Disorder of Consciousness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Louis De Beaumont, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-2279
Record Dates: First submitted 2023-03-20; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Brain Injury Traumatic Severe; Disorder of Consciousness; Brain Injuries
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-Hz tACS Stimulation Group (Active Comparator): tACS stimulation will be delivered over to parieto-occipital sites using only 2-minute ramp up and down and a continuous 20-minute 10 Hz sinusoidal current administered. The stimulation electrode montage will be identical for both conditions.
  Interventions: Device: Active Transcranial alternative current stimulation
- Sham Stimulation Group (Sham Comparator): Sham stimulation will be delivered over to parieto-occipital sites using only 2-minute ramp up and down, without any sinusoidal current administered for 20 minutes. The stimulation electrode montage will be identical for both conditions.
  Interventions: Device: SHAM Transcranial alternative current stimulation

INTERVENTIONS:
Device: Active Transcranial alternative current stimulation — GTEN 200 (Magstim-EGI, OREGON, USA). The current will be administered via an amplifier connected to an EEG system of 128-Channel Geodesic Sensor Net (Magstim-EGI, Oregon, USA) with sponge-based electrode nets.
  tACS stimulation will be applied for 20 minutes for 5 consecutive days via a bilateral electrode montage of 5 electrodes per hemisphere over parieto-occipital cortical sites. Specific stimulation electrodes for both conditions will be: [right hemisphere: E83, E90, E96, E84, E91] and for the [left hemisphere: E58, E65, E70, E66, E59]. The intensity of the applied alternative current (AC) will be a maximum of 1 mA peak-to-peak. The stimulation frequency will be adjusted to 10 Hz (median value of the alpha frequency band) for the tACS condition.
  Arms: 10-Hz tACS Stimulation Group
Device: SHAM Transcranial alternative current stimulation — GTEN 200 (Magstim-EGI, OREGON, USA). The current will be administered via an amplifier connected to an EEG system of 128-Channel Geodesic Sensor Net (Magstim-EGI, Oregon, USA) with sponge-based electrode nets.
  SHAM stimulation will be applied for a 2-minute ramp-up, then the current will stop for 20 minutes, followed by a 2-minute ramp-down. This will be applied for 5 consecutive days via a bilateral electrode montage of 5 electrodes per hemisphere over parieto-occipital cortical sites. Specific stimulation electrodes for both conditions will be: [right hemisphere: E83, E90, E96, E84, E91] and for the [left hemisphere: E58, E65, E70, E66, E59]. The intensity of the applied alternative current (AC) will be a maximum of 1 mA peak-to-peak. The stimulation frequency will be adjusted to 10 Hz (median value of the alpha frequency band) for the ramp-up and down in the SHAM conditions.
  Arms: Sham Stimulation Group

SUMMARY:
This study first aims to validate the feasibility of a multimodal 5-day 20-minute tACS protocol in subacute brain-injured patients with a disorder of consciousness during their ICU stay, and conduct a clinical pilot study (validation phase). Upon completion of this validation phase and according to obtained results, a randomized clinical trial will be conducted to compare the effects of the 5-day active 10Hz-tACS protocol with a 5-day sham-tACS protocol on brain dynamics modulation. This study will also compare intervention conditions on recovery of consciousness, cognition and function using short-term and long-term measurements.

DETAILED DESCRIPTION:
Background: After a severe brain injury, a significant number of patients remain in a state of altered consciousness and the outcome remains difficult to prognosticate. There is a lack of evidence-based therapeutic interventions available for patients with disorders of consciousness; some evidence has been gathered for non-invasive brain stimulation, but these have targeted chronic patients. The objective of the validation phase will be to evaluate the differential feasibility parameters of conducting a 5-day tACS stimulation protocol in the ICU and the quality of data collection according to the various measurement modalities, to establish requirements to be used in a larger-scale study. This phase will also implicate a clinical pilot to confirm and assess the effect size of the primary outcome and sample size requirements for a clinical trial. Following completion, a clinical trial will be conducted to evaluate short-term and long-term neurophysiological effects of an optimized, multi-session tACS intervention in subacute brain-injured patients on their consciousness and functional recovery (as measured by complementary behavioural/functional scales), related brain oscillations and network dynamics.

Validation phase: In addition to conducting the following methods and design protocol, these measures will be acquired during the validation phase to assess the feasibility of this single-site study.

Recruitment rate and retention: Estimated number of patients in this condition in this ICU per year, estimated patient survival rates, number of eligible patients over a 12-month recruitment period; percentage of patients recruited, attrition, presence of competitive studies, etiologies and compliance of the families through experimental protocol and longitudinal assessment (12-month period).

Site demographics: Personnel's availabilities, Availability/accessibility of study coordinators, technicians, doctors and nurses; competency of the experimental team to conduct the experimental protocol.

Site infrastructure: Material storage (biological samples (centrifuge, freezer), Material obtention (Lidocaine obtention and renewal; EEG equipment), Data storage (clinically secure on-site servers).

Investigators' team requirements: Personnel requirements and the number of personnel required for the protocol's conductance.

Assessing the investigator's readiness in terms of standard care (eligibility decisions according to clinical profiles ), targeted study population and population recruited, and familiarity with the use of tools and technology.

Acceptability within the clinical care team's ecosystem: document pitfalls, difficulties and requirements to facilitate the clinical care team's adherence Quality of data collection: quality of EEG signal data in different clinical settings across main acquisition hospital sites; percentage of data acquisition completion; encountered data acquisition obstacles; assessment the estimated acquisition time for each measure and actual measuring times.

Methods/design:

The investigators will recruit brain-injured patients traumatic and non-traumatic etiologies (e.g., traumatic brain injury, anoxic brain injury, subarachnoid hemorrhage). Twelve patients will be recruited for the validation phase. The sample size estimation for the clinical trial based on a Student's t-test is 138 (2 groups of 69 patients) to reach a power of 80% to detect a statistically significant difference in the amplitude of alpha activity between active and sham groups, assuming a dropout/death rate of 20% and a significance level of 5%. These parameters are calculated according to a randomized, sham-controlled clinical trial comparing a 4-week tDCS protocol on patients with disorders of consciousness. The main outcome was a behavioral assessment, whereas this study's main outcome is neurophysiological, which is more sensitive to detect modulation effects. Additionally, this estimate will be readjusted according to the clinical pilot's results.

The study protocol will be activated once the medical team states clinical stability for the patients and withdrawal of continuous sedation has surpassed a minimum of 24 hours, without recovery of responsiveness.

Patients will participate in 7 consecutive experimental days including :

Day 0: Baseline measurements: Blood samples ( pharmacological agents dosage, the plasma expression of glial fibrillary acidic protein (GFAP) and isolation of exosomes derived from neurons (EDNs), astrocytes (EDAs) and microglia (EDMs)), Behavioral outcomes (Coma Recovery Scale-Revised (CRS-R), Glasgow Coma Scale (GCS) and Full Outline of Unresponsiveness (FOUR) Score) will be additionally measured for Unresponsive Wakefulness patients), pupillometry (photo motor reflex), and actigraph installation.

Days 1 to 5 (the following sequential procedure):

CRS-R/FOUR/GCS Pupillometry (PLR) 5-minute resting-state EEG 20-minute tACS/sham 5-minute resting-state EEG Pupillometry (PLR) CRS-R

5-minute resting-state 60-minute post-tACS condition/sham condition

5-minute resting-state 120-minute post-tACS condition/sham condition

Day 6:

CRS-R Pupillometry (PLR) 5-minute resting-state EEG

Day 7: After an interval of one-week post-5-day tACS/sham protocol, the following measurements will be acquired: CRS-R, Pupillometry (photo motor reflex), and 5-minute resting-state EEG. The actigraph will be withdrawn the during this same session.

At 3,6 and 12 months post-tACS, phone assessments will be conducted to measure long-term functional recovery using the following tools: Glasgow Outcome Scale- Extended, Disability Rating Scale, Functional Independence Measure and Burden Scale for Family Caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old; Glasgow Coma Scale score remaining ≤ 12 following a minimum of 24 hours after the withdrawal of continuous sedation (if applicable).
* The included brain injury etiologies for the Unresponsive Wakefulness Syndrome(UWS) or Minimally Conscious State (MCS) are traumatic and non-traumatic (e.g., traumatic brain injury, anoxic brain injury, subarachnoid hemorrhage).

Exclusion Criteria:

* Focal brain lesion(s) in the occipital and parietal lobes located at stimulation site
* Pre-existing severe neurological conditions/disorders involving cognitive deficits such as neurodegenerative diseases (ALS, dementia, Parkinson's), hereditary conditions (e.g. Huntington's Chorea), CNS disorders (previous moderate-severe CBT)
* History of epilepsy (patient with a seizure episode in response to non-exclusive active tACS intervention)
* Aneurysm clip(s), subdural brain electrodes, metallic brain, an implant, implantable neurostimulator
* Craniectomy with no bone flap
* Cervical collar limiting access to the occipital region
* Participation in a current (or previous) study that may have a confounding effect, as assessed by the research team.

To facilitate recruitment, upon medical consent family members of patients who present inclusion criteria before meeting the protocol activation criteria will be approached by the research team to get informed consent. The study will be activated once the medical team confirms clinical stability and withdrawal of continuous sedation for a minimum of 24 hours. The study protocol will not be activated if there is: Constant and intense agitation at the time of study activation, the presence of invasive neurological monitoring (ICP and/or PbtO2), GCS > 12 after 24 hours of continuous sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Single-site recruitment rates | 1 year
  Quantify the frequency of recruitment in the entire study's protocol for the specific population in the Intensive Care Unit.
Retention rates | over the 2-week course of the experimental protocol and at 3, 6 and 12 month time points
  Assess completion and participation in the entire study's from participants and their caregivers; for the intervention protocol as well as for longitudinal measures over time [3,6,12 months]
Change in EEG spectral power of the alpha band activity | It will be measured over the 2-week course of the experimental protocol
  EEG measures cortical electrical activity. Increase in the alpha band spectral power after the end of the 5-day 20-minute 10 Hz tACS intervention would indicate the specificity of the modulation's effect.
Change in Functional Connectivity based on EEG signal | It will be measured over the 2-week course of the experimental protocol
  Examine changes in the statistical relationship between specific electrophysiological signal parameters in time.

SECONDARY OUTCOMES:
Changes in Coma Recovery Scale Revised (CRS-R) score throughout the protocol. | It will be measured over the 2-week course of the experimental protocol
  The Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioural assessment of consciousness. It contains 23 items hierarchically presented and divided into 6 sub-scales (auditory, visual, motor, oro-motor/verbal, communication and arousal). The score is based on the presence or absence of behaviours in response to sensory stimulations. The best-observed response in each sub-scale is used to differentiate between the level of consciousness [Unresponsive Wakefulness Syndrome patients (UWS), minimally conscious state (MCS- and MCS +) and emergence (EMCS)]. The diagnosis is obtained from the quality of observed behaviours (e.g., the ability of visual tracking means that the patient is minimally conscious). The total score ranges between 0 and 23. Baseline measures [Day 0], daily measures [Day 1 to 5: Pre and post-tACS/sham] and up to a week after the protocol [Day 6: 24-hour after the 5-day protocol (post-24) and a week post the 5-day protocol (Day 7)].

OTHER OUTCOMES:
Monitor non-invasively changes in the pupillary light reflex across the protocol | It will be measured over the 2-week course of the experimental protocol
  Pupillary dilation is usually associated with a behavioural change to a more active state.
Monitor the recovery of wake-sleep cycles across the protocol | It will be measured over the 2-week course of the experimental protocol
  Recovery from disorders of consciousness among moderate to severe TBI patients has been linked to a recovery in the consolidation of the 24-hour wake-sleep cycle when measured by an actigraphy device.
Characterize pharmacological agents, dosage of the plasma expression of the glial fibrillary acidic protein (GFAP) and to isolate exosomes derived from neurons (EDNs), astrocytes (EDAs) and microglia (EDMs). | Baseline measure (day 0)
  Initial blood sample analyses
Longitudinal changes on global outcomes using GOSE and CPCs between conditions tACS and sham at 3, 6 and 12 months post-completion of the experimental protocol. | 1 year
  The Glasgow Outcome Scale-Extended (GOSE) assesses the overall outcome of patients that suffered from a Traumatic Brain Injury. This scale is used to categorize patients into 5 main categories and 3 subdivisions (Lower and Upper).The Cerebral Performance Category (CPC) score is widely used in research to assess neurological outcomes following cardiac arrest. This scale ranges from 1 (good) to 5 (poor) neurological outcomes.
Longitudinal changes on Disability Rating Scale (DRS) and Functional Independence Measure (FIM) between conditions tACS and sham at 3, 6 and 12 months post-completion of the experimental protocol. | 1 year
  Complementary measures to assess functional recovery outcomes. The DRS assesses functional recovery. It contains 8 items and the maximal score a patient can obtain is 29. The FIM assesses the functional status of a patient based on the level of assistance required based on 6 areas of function. Each item is scored on a 7-point ordinal scale.
Changes in Subjective Burden Scale for Family Caregivers (BSFC-s) between conditions tACS and sham at 3, 6 and 12 months post-completion of the experimental protocol. | 1 year
  The BSFC-s assesses the perceived burden of caregivers. This instrument includes 10 items each including a 4-point scales statements.
Changes in perceived health-related quality of life using EQ-5D-L5 between conditions tACS and sham at 3, 6 and 12 months post-completion of the experimental protocol. | 1 year
  The EQ-5D-5L is a self-assessed, health-related quality-of-life questionnaire. This scale includes 5-components : mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Martens G, Lejeune N, O'Brien AT, Fregni F, Martial C, Wannez S, Laureys S, Thibaut A. Randomized controlled trial of home-based 4-week tDCS in chronic minimally conscious state. Brain Stimul. 2018 Sep-Oct;11(5):982-990. doi: 10.1016/j.brs.2018.04.021. Epub 2018 May 2. PMID 29759943
- [Derived] De Koninck BP, Brazeau D, Deshaies AA, Briand MM, Maschke C, Williams V, Arbour C, Williamson D, Duclos C, Bernard F, Blain-Moraes S, De Beaumont L. Modulation of brain activity in brain-injured patients with a disorder of consciousness in intensive care with repeated 10-Hz transcranial alternating current stimulation (tACS): a randomised controlled trial protocol. BMJ Open. 2024 Jul 11;14(7):e078281. doi: 10.1136/bmjopen-2023-078281. PMID 38991682